CLINICAL TRIAL: NCT01481077
Title: PPL GLAU 13: A Randomized Phase 2 Study of the Effect of Plug Placement on Efficacy and Safety of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Dose Evaluation Study of the Effect of Plug Placement on the Efficacy and Safety of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 13
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension (OH)
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Latanoprost-PPDS
- Treatment B (Experimental)
  Interventions: Drug: Latanoprost-PPDS
- Treatment C (Experimental)
  Interventions: Drug: Latanoprost-PPDS

INTERVENTIONS:
Drug: Latanoprost-PPDS — Sustained release for 12 weeks

SUMMARY:
The purpose of this study is to determine the effect of plug placement on the efficacy, safety and duration of effect of the L-PPDS (latanoprost punctal plug delivery system).

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Diagnosis of bilateral open angle glaucoma or ocular hypertension
* Unmedicated IOP must be ≥22mm Hg

Exclusion Criteria:

* Any significant vision loss in the last year
* No contact lens use for the length of the study
* Abnormal eye lids, eye infection or diseases to the eye
* Recent eye surgery
* Uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 12 weeks to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Cadden, Study Director — QLT Inc.
Locations (11):
- United States (11):
  - Vold Vision, Springdale, Arkansas
  - Glaucoma Consultants of Colorado, PC, Denver, Colorado
  - Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - Ophthalmology Consultants Inc., Des Peres, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd, Washington, Missouri
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Abrams Eye Institute, Las Vegas, Nevada
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - University Eye Surgeons, Maryville, Tennessee
  - Total Eye Care, P.A., Memphis, Tennessee